CLINICAL TRIAL: NCT00724360
Title: A Phase II Trial Evaluating the Safety and the Efficacy of Trastuzumab in Relapsed/Refractory HER2 Positive B-acute Lymphoblastic Leukemia Patients.
Brief Title: Trastuzumab for HER2 Positive Relapsed/Refractory B-Acute Lymphoblastic Leukemia (B-ALL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD04/2-T
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Relapsed/Refractory Leukemia
Keywords: relapsed/refractory; HER2; positive; B-ALL; trastuzumab
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Trastuzumab

INTERVENTIONS:
Drug: Herceptin (trastuzumab) — Administered as a 4 mg/kg intravenous loading dose followed by 2 mg/kg weekly for at least 2 months and/or until progression

SUMMARY:
This is a multicenter open-label phase II trial of trastuzumab in patients with HER2 positive B-ALL in relapse, or with refractory disease. Herceptin is administered as a 4 mg/kg intravenous loading dose followed by 2 mg/kg weekly for at least 2 months and/or till progression. Response and HER2 expression are assessed each month by bone marrow aspirate.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* B-ALL in relapse
* refractory B-ALL-performance status of 0-2 on the Eastern Cooperative Oncology Group scale
* adequate hepatic and renal functions (AST or ALT <= 5 times the upper limit of normal creatinine < 2 times the upper limit of normal)
* > 20% blasts in bone marrow,
* > 30% of bone marrow blast population HER2 positive as assessed by immunophenotyping

Exclusion Criteria:

* Previous treatment by trastuzumab
* FEVG < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-11; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Response rate: Response was defined either as complete response (CR), CR without recovery of platelet (CRp), or partial response (PR)

SECONDARY OUTCOMES:
Trastuzumab efficiency concerning transfusional needs
Overall survival
Leukemia free survival
cytogenetic response rate
Trastuzumab tolerance profile

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Mondor Hospital, Créteil
  - Grenoble Hospital, Grenoble
  - Institut Paoli Calmettes, Marseille
  - CHU, Nantes
  - St Louis Hospital, Paris
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg

REFERENCES:
- [Derived] Chevallier P, Robillard N, Charbonnier A, Raffoux E, Maury S, Carras S, Chabrot C, Fohrer C, Bernard M, Blade JS, Etienne A, Talmant P, Delaunay J, Guillaume T, Mohty M, Bene MC, Ifrah N, Dombret H. Trastuzumab for treatment of refractory/relapsed HER2-positive adult B-ALL: results of a phase 2 GRAALL study. Blood. 2012 Mar 15;119(11):2474-7. doi: 10.1182/blood-2011-11-390781. Epub 2012 Jan 20. PMID 22267607